CLINICAL TRIAL: NCT01790685
Title: Ozurdex for Retinal Vein Occlusion Study (ORVO Study)
Acronym: ORVO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Peter A Campochiaro, MD, MD, Johns Hopkins University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00079951
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Results first posted 2015-04-03 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRVO (Other): Central Retinal Vein Occlusion
  Interventions: Drug: dexamethasone implant
- BRVO (Other): Branch Retinal Vein Occlusion
  Interventions: Drug: dexamethasone implant

INTERVENTIONS:
Drug: dexamethasone implant
  Other Names: Ozurdex

SUMMARY:
To measure the pro-permeability factors in the aqueous humor of patients with persistent/recurrent macular edema after an injection of Ozurdex.

DETAILED DESCRIPTION:
To measure various pro-permeability factors in the aqueous humor of patients with persistent/recurrent macular edema despite prior treatment with anti-VEGF agents at baseline and at 4 weeks after intraocular injection of OZURDEX.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age more than or equal to 18 years
* Diagnosis of macular edema due to central or branch retinal vein occlusion
* Intraretinal or subretinal fluid in the macula determined by Spectralis OCT
* Best corrected visual acuity score in the study eye of 20/30 to 20/400 inclusive (Snellen equivalents using the ETDRS protocol at a distance of 4 meters)
* In the opinion of the investigator, decreased vision in the study eye is due to foveal thickening from vein occlusion and not from other obvious causes of decreased vision
* Persistent or recurrent edema despite prolonged treatment with an anti-VEFG agent

Exclusion Criteria:

* Scatter laser photocoagulation or macular photocoagulation within 3 months of study entry in the study eye
* Intraocular surgery in the study eye within 3 months of study entry
* Use of intraocular or periocular injection of steroids in the study eye (e.g., triamcinolone) within 4 months of study entry
* Previous use of an anti-VEGF drug within 1 month of study entry
* Yttrium-Aluminum-Garnet (YAG) laser capsulotomy within 1 month of study entry
* Any condition that the investigator believes would pose a significant hazard to the subject if investigational therapy were initiated.
* Inability to comply with study or follow up procedures
* History of glaucoma or documented history of steroid-induced glaucoma.
* Patients with active or suspected ocular or periocular infection, including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
* Aphakic eyes with rupture of the posterior lens capsule.
* Eyes with ACIOL and rupture of the posterior lens capsule.
* Patients with hypersensitivity to dexamethasone or to any other components of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 patients from the clinic population of the Wilmer Eye Institute were recruited,
Groups:
- CRVO: Central Retinal Vein Occlusion
  dexamethasone implant
- BRVO: Branch Retinal Vein Occlusion
  dexamethasone implant
Period: Overall Study
Arm/Group | CRVO | BRVO
Started | 23 | 17
Completed | 23 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRVO | BRVO | Total
Number analyzed (Participants) | 23 | 17 | 40
Age, Continuous [Median (Full Range); unit: years] | 74 [54 to 90] | 72 [54 to 89] | 73 [54 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had a >30% Decrease in the Aqueous Levels of Various Vasoactive Proteins 4 Weeks After an Injection of Ozurdex
Description: Vasoactive protein arrays and Enzyme linked immunosorbent assays were done for patients at baseline and week 4 visit to measure the levels of various pro-permeability factors including VEGF, SDF-1 and Angiopoietin-2.
Time Frame: 4 months
Population: All enrolled (23 CRVO and 17 BRVO) patients completed the study. All patients were injected with Ozurdex, however microarrays were run on only 11 CRVO and 17 BRVO patient samples. Microarray data from 11 CRVO and 11 BRVO patients was analyzed.
Measure: Number; unit: participants
Arm/Group | CRVO | BRVO
Number analyzed (Participants) | 11 | 11
participants
  HGF | 7 | 5
  EG-VEGF | 7 | 4
  Activin-A | 4 | 6
  IGFBP-1 | 7 | 4
  IGFBP-2 | 7 | 6
  IGF-BP3 | 7 | 6
  Endostatin | 7 | 6

ADVERSE EVENTS:
Arm/Group | CRVO | BRVO
Serious Adverse Events (participants affected / at risk) | 1/23 | 2/17
Other Adverse Events (participants affected / at risk) | 8/23 | 5/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRVO (N=23) | BRVO (N=17)
Patient fell down the stairs and was hospitalized for a cerebral bleed. (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
The patient was hospitalized for an infection (Infections and infestations) | 0 (0) | 1 (1)
Patient fell and hit head on the back of a chair resulting in trauma and infection in the study eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
The patient was hospitalized for stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRVO (N=23) | BRVO (N=17)
Increase in IOP in study eye (Eye disorders) | 3 (3) | 3 (3)
Redness of study eye after drug injection (Eye disorders) | 2 (2) | 2 (2)
Patient had an uneventful fall (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is a restriction on the PI regarding disclosure of study results, which will be updated once the manuscript is published.